CLINICAL TRIAL: NCT04281043
Title: Quality of Life After Robotic Surgery as Primary Treatment for Endometrial Cancer
Brief Title: Quality of Life After Robotic Surgery for Endometrial Cancer
Acronym: QoL
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Hjalmar Svensson Foundation (Unknown); Assar Gabrielsson Foundation (Unknown); Göteborg Medical Society (Unknown)
Responsible Party: Principal Investigator, Anna Lindfors, Medical Doctor, Sahlgrenska University Hospital
Other Study IDs: QoL Robot
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Quality of Life; Endometrial Cancer; Surgery--Complications; Gynecologic Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate how robotic assisted laparoscopic surgery affects the quality of life of women who are treated with primary surgery for endometrial cancer. So far, very little has been published and basically no long-term follow-up.

Included patients respond to questionnaires preoperatively, 2 weeks after surgery and 3 months and 12 months after surgery.

Each patient thus answers the questionnaires (the same) on four occasions. The questionnaires used are validated and used extensively internationally. The first survey has two parts, QLQ30 and the module for endometrial cancer EN24. In addition the study includes use PHQ -9 and GAD 7.

DETAILED DESCRIPTION:
Objective: In a pilot study to prospectively analyze the quality of life using QLQ-C30, EN-24, PHQ-9 and GAD7 in women undergoing primary surgery with robotic assisted laparoscopy for corpus cancer before and up to one year after surgery.

The study aims to describe how, to what extent and when in relation to primary surgery women's quality of life is affected after the diagnosis of endometrial cancer. The long-term goal of the work is to be able to deploy any resources if needs exist, and in this case at a time when they are most useful, to promote the quality of life of the affected women.

Question: How and when is the quality of life of women undergoing surgery for endometrial cancer affected? Is there any particular area / domain that is affected more than others and is this impact persistent over time? Method: The international and validated survey, QLQ-C30 with the addition of EN24, developed by the European Organization for Research and Treatment of Cancer (EORTC) for quality of life measurement specifically for endometrial cancer in addition to PHQ-9 and GAD7 to evaluate depression and anxiety symtoms, is planned to be used just before primary surgery, 1-2 weeks, 3 months and 1 years postoperatively.

Referens to the QLQ30 questionnaire below.

Patients are included at Department of Obstetrics and Gynecology, Sahlgrenska University Hospital, Gothenburg, Sweden for one year.

All patients included should give their oral and written consent. All data will be registered coded and analyzed without personal identification number according to the scoring manual from EORTC.

Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JCJM, Kaasa S, Klee MC, Osoba D, Razavi D, Rofe PB, Schraub S, Sneeuw KCA, Sullivan M, Takeda F.

The European Organisation for Research and Treatment of Cancer QLQ-C30: A quality-of-life instrument for use in international clinical trials in oncology. Journal of the National Cancer Institute 1993; 85: 365-376.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years of age
* scheduled for primary surgery for histologically verified endometrial cancer (regardless of histological type or degree),
* tumor clinically restricted to the uterus (presumptive FIGO stage I or II),
* speaks and reads Swedish,
* capable of completing the questionnaire independently.

Exclusion Criteria:

* Clinical or radiological cancer outside the uterus
* preoperative radio / chemotherapy.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients planned for primary surgery with robotic technique for endometrial cancer at Department of Obstetrics and Gynecology, Sahlgrenska University Hospital, Gothenburg, Sweden will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life at 3 months | 3 months
  Quality of Life at 3 months postoperatively compared to preoperatively The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  Allofthescalesandsingle-itemmeasuresrangeinscorefrom0to100. Ahighscalescore represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  The attached module EN24 has 3 functional scales and several symptom scales, which scores follows the same system.
Quality of Life at 12 months | 12 months
  Quality of Life at 12 months postoperatively compared to preoperatively The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  Allofthescalesandsingle-itemmeasuresrangeinscorefrom0to100. Ahighscalescore represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  The attached module EN24 has 3 functional scales and several symptom scales, which scores follows the same system.

SECONDARY OUTCOMES:
Anxiety scores | 3 months
  Scores on GAD7 3 months postoperatively compared to preoperatively Scores 0-21, were a higher scores is associated with more symptoms.
Anxiety scores | 12 months
  Scores on GAD7 12 months postoperatively compared to preoperatively
Depression scores | 3 months
  Scores on PHQ9 3 months postoperatively compared to preoperatively. Scores 0-27 were a high score is associated with more symptoms.
Depression scores | 12 months
  Scores on PHQ9 12 months postoperatively compared to preoperatively. Scores 0-27 were a high score is associated with more symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- 1Department of Obstetrics and Gynecology, Sahlgrenska University Hospital, Gothenburg, Sweden, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided